CLINICAL TRIAL: NCT07391384
Title: Evaluation of the Effect of Thymoquinone Hydrogel With Bone Graft in Comparison to Bone Graft Only Around Immediate Implant (Randomized Controlled Clinical Trials)
Brief Title: Thymoquinone Around Immediate Implant
Acronym: Thymoquinone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: shaimaa hamdy (Other)
Responsible Party: Sponsor-Investigator, shaimaa hamdy, lecturer of periodontology, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Thymoquinon+ immediate implant; committee 1238 (Other: ethical committee faculty of dentistry minia university)
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Immediate Dental Implant Placement; Jumping Gap; Primary Stability of the Implants
Keywords: immediate implant; thymoquinone; hydrogel; bone graft
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study will include 44 immediate implants replacing non-restorable posterior teeth. The patients were randomly assigned in equal numbers to two groups using http://www.randomizer.org Group I (Control): 22 implants will be inserted immediately after tooth extraction with xenograft.
  Group II (Study): 22 implants will be inserted immediately after tooth extraction, combined with xenograft and TQ gel.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All participants, investigators, surgeons, and outcomes investigator are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- surgical implants will inserted immediately after teeth extraction with xenograft. (Placebo Comparator): immediat implant placement with bone graft hydrogel
  Interventions: Procedure: group 1 xenograft hydrogel
- study group (Active Comparator): surgical placement of 22 implants will inserted immediately after teeth extraction, combined xenograft and TQ gel.
  Interventions: Procedure: immediat implant placement wit TQ and bone graft hydrogel placement around implant

INTERVENTIONS:
Procedure: group 1 xenograft hydrogel — 22 implants will inserted immediately after teeth extraction with xenograft.
  Other Names: control group
  Arms: surgical implants will inserted immediately after teeth extraction with xenograft.
Procedure: immediat implant placement wit TQ and bone graft hydrogel placement around implant — 22 implants will inserted immediately after teeth extraction, combined xenograft and TQ gel.
  Arms: study group

SUMMARY:
use of Thymoquinone hydrogel with bone graft in comparison to bone graft only around immediate implant-this hydrogel fill the jumping zone in comparison to using hydrogel bone graft only to increase primary stability and enhance osseointegration

DETAILED DESCRIPTION:
Immediate dental implant placement has gained popularity for replacing extracted teeth due to its advantages, including shorter treatment time, better preservation of alveolar bone volume, and enhanced aesthetic outcomes. However, the success of immediate implants largely relies on achieving optimal osseointegration, defined as the direct structural and functional bond between living bone and the surface of a load-bearing implant. Factors such as implant surface properties, surgical techniques, and patient-specific variables, including bone quality, influence this process.

Extensive research has aimed to enhance bone-to-implant contact (BIC), a key factor for successful osseointegration. Strategies include modifying implant surface morphology and applying bioactive agents, both intended to improve BIC and support long-term implant integration.

Many preclinical and clinical studies have documented the regeneration of horizontal gaps smaller than 2 mm in the presence of a stable blood clot but when the peri-implant gap distance was more than 2mm the bone graft should be used to seal this bony defect.

Herbal medicine has gained researchers' attention for the treatment of oral and periodontal diseases due to its beneficial, safer, integrated effects, reduced cost an minimal side effects.Nigella sativa (NS) is known as "black seed", a flower in plant that grows in Middle East, some Asian and Mediterranean countries.

Thymoquinone (TQ) is one of the main bioactive components of NS, it has valuable therapeutic effect because of its anti-oxidant, antimicrobial, analgesic, anti-inflammatory, antihypertensive, anti-histaminic, hypoglycemic, hepatoprotective, anticarcinogenic, and immune-activating properties. Considering the anti-inflammatory, antimicrobial and antioxidant characteristics of TQ, it may play a significant role in preventing the initiation, progression and treatment of periodontal diseases.

NS and its active ingredient TQ has been used for the treatment of hypertension, cancer, rheumatoid arthritis, diabetes, bronchial asthma, hypertension, obesity, Behcet's disease, liver damage and other metabolic and autoimmune disorders. TQ was found to be responsible for the therapeutic effect of NS.

NS and TQ displayed abundant therapeutic properties on different oral diseases and conditions such as dental caries, intracanal medication, oral ulcerations, mucositis, wound healing, postextraction bone healing, oral cancer, gingival and periodontal diseases. The effects of TQ in periodontal disease-associated settings and their modes of action with potential benefits for periodontal therapy have been investigated in several studies. These include in vitro studies, in vivo (animal) studies, and clinical studies (RCTs).

The mode of action of TQ in periodontal diseases is anti-inflammatory and anti-oxidant activity through suppression of inflammatory cytokines (IL-1b,IL-6,TNF-ἀ, PGE), Activation of IL-10 and suppression of NO. The anti-bacterial properities through suppression of bacterial resistance and Disintegration of bacterial membranes. Stem cell modulatory effect through activation of stem cell migration and stem cell immunomodulation and potentially regenerative mechanisms of these rich natural compounds.

Different studies evaluated the effect of different gel materials around immediate implant placement such as melatonin and hyalourinic acid gels, topical Vit.D around immediate implant and simvastatin gel .

To our knowledge, there is no human study that evaluate the effect of TQ in management of gap distance around immediate implant placement. Therefore, the aim of the present study was to evaluate the effect of topically TQ gel around immediate implants placement both clinically and radiographically.

Aim of the study Primary outcome: Evaluate the effect of TQ hydrogel around immediate implant placement clinically and radiographically.

Secondary outcome: To Compare The effect of TQ hydrogel with bone graft in comparison to bone graft only around implant clinically and radiographically.

.

Patients and Methods

Study design:

This Randomized controlled clinical trials will be conducted on 44 patients. The entire patients will be selected from the out patients clinic of the Oral Medicine, Oral Diagnosis, and Periodontology Department. Faculty of Dentistry, Minia University.

Sample size calculation:

The sample size was calculated using G*Power (version 3.1.9.7) for an ANCOVA (fixed effects, including main effects and interactions) that compares two groups while adjusting for one covariate. Assuming an effect size of f = 0.56 (partial), with a two-group design, an alpha level (α) of 0.05, and a power (1-β) of 0.95, the required total sample size is 44 participants, which breaks down to 22 participants per group. With this sample size, the denominator degrees of freedom would be 41 (calculated as total N, number of groups, number of covariates: 44 - 2 - 1 = 41). This setup allows for sufficient power to detect an effect while accounting for the covariate.

The complete treatment plan will be explained to all patients including detailed steps, risks, and expected results and their full signed consent will be obtained prior to entry into the study. The study will be complied with the rules set by the International Conference on Harmonization Good Clinical Practice Guidelines, and the Declaration of Helsinki and the research ethics committee of the Faculty of Dentistry, Minia University.

Study groups and randomization The study will include 44 immediate implants replacing non-restorable posterior teeth. The patients were randomly assigned in equal numbers to two groups using http://www.randomizer.org Group I (Control): 22 implants will inserted immediately after teeth extraction with xenograft.

Group II (Study): 22 implants will inserted immediately after teeth extraction, combined xenograft and TQ gel.

Preoperative phase Clinical examination Personal data, including name, age, gender, occupation and contact information, will be collected for each patient.

A detailed medical and dental history will be taken to exclude those with conditions or habits that could negatively impact implant stability.

Oral hygiene will be assessed and patients will refer to the Oral Medicine and Periodontology Department for scaling and polishing. Occlusion will be evaluated to ensure proper alignment and contact.

The surgical procedure and potential complications (e.g., bleeding, pain, swelling, implant failure) will be explained to each patient. Photographs and follow-up X-rays will be used for documentation and monitoring healing. These data will be collected to ensure each patient will meet the inclusion criteria.

Preparation of TQ gel:

TQ-loaded niosomes will be prepared using the ethanol injection method (Mostafa et. al.). The formulation consisted of Span 60, cholesterol, PEG 4000, and TQ in a weight ratio of 90:35:5:10, respectively. For a representative batch, 90 mg of Span 60, 35 mg of cholesterol, 5 mg of PEG 4000, and 20 mg of TQ will be used. Span 60 and cholesterol will be dissolved in 5 mL of absolute ethanol (organic phase) and gently heated in a water bath at 60-70 °C with stirring until a clear solution will be obtained. Meanwhile, PEG 4000 will be dissolved in 10 mL of preheated phosphate-buffered saline (PBS, pH 7.4) to prepare the aqueous phase, which will be maintained at the same temperature as the organic phase.

The ethanolic lipid solution will be injected slowly into the aqueous phase at a rate of approximately 0.5-1 mL per minute under continuous magnetic stirring (800 rpm) while maintaining the temperature at 60-70 °C. Stirring will continued for an additional 20 minutes after the injection will completed to ensure proper vesicle formation. The residual ethanol will then removed by rotary evaporation under reduced pressure until negligible solvent remained. The resulting niosomal dispersion will then sonicated in an ice bath using a water bath sonicator for 2 min to reduce particle size and achieve uniform distribution. Thymoquinone will encapsulated into the niosomes using post insetion approach. In brief, TQ (20 mg) will dissolved into 2 ml of ethanol and added to the preformed niosomal suspension under stirring and incubated for 2 hr at 37 °C.

Unencapsulated thymoquinone will separated by ultracentrifugation at 15000 rpm for 60 minutes at 4 °C, and the collected niosomal pellet will resuspended in PBS to the original volume. The purified thymoquinone niosomes will stored at 4 °C, protected from light, until further characterization.

The encapsulation efficiency (EE%) was determined by quantifying the amount of free thymoquinone in the supernatant after purification using a validated UV-VIS method. The detection wavelength will set at 254 nm. The EE% will calculated using the equation EE% = [(Wt - Wf) / Wt] × 100, where Wt is the total thymoquinone added and Wf is the amount of free drug detected in the supernatant.

The prepared niosomes will characterized for their mean particle size, polydispersity index (PDI), and zeta potential using dynamic and electrophoretic light scattering techniques (DLS/ELS) at 25 °C. Samples were diluted 20-100-fold in PBS before measurement. Each measurement will performed in triplicate, and results will expressed as mean ± SD. The surface morphology of the niosomes will examined by scanning electron microscopy (SEM). A drop of diluted niosomal dispersion wil placed on an aluminum stub, air-dried under vacuum, sputter-coated with a thin layer of gold-palladium (≈5 nm), and imaged at an accelerating voltage of 5-15 kV.

The light-stability study will conducted to evaluate the photostability of TQ within the niosomal system. Aliquots of free drug and niosomal dispersion (5 mL each) will stored in clear glass vials exposed to UV light at 25 ± 2 °C, and analyses will performed at predetermined time intervals for drug content. The percentage of TQ remaining will plotted against time to assess photostability of the niosomes.

Surgical phase:

1. The surgical procedures, will be carried out following strict infection control protocols. Patients will be instructed to rinse with 0.1% chlorhexidine (Hexitol antiseptic mouthwash, Arabian Drug Company (ADCO), Cairo, Egypt) and the peri-oral tissues will be disinfected with povidone-iodine (Betadine, Nile Co. for Pharma, Cairo, Egypt).
2. Local anesthesia will be injected via the infiltration or nerve block technique using 4% articaine hydrochloride with 1:100,000 epinephrine (Artinibsa, Inibsa Dental SLU, Spain).
3. Atraumatic tooth extractions will be performed, preserving the alveolar bone. The dimensions of the extraction socket and residual bone will be evaluated using a periodontal probe, in addition to measuring the width and length of the extracted tooth root, to ensure appropriate implant selection. Measurements will be taken to confirm compatibility with the planned implant size and ensure proper placement.
4. Osteotomy drilling followed a standardized protocol, using sequential drills and adequate torque and speed under copious irrigation.
5. In the control group, xenograft will be applied to both the implant surface and the osteotomy site after implant placement.

While in study group, xenograft mixed with TQ gel will be inserted around implant.

Post-surgical phase:- Post-surgical instructions Following surgery, patients will receive detailed postoperative care instructions and prescribed medications including Cataflam 50 mg tablets (Diclofenac potassium) a non-steroidal anti-inflammatory drug taken twice daily for 4 days and Hexitol mouth wash (Chlorhexidine HCL 0.12%) an antiseptic mouth wash used twice daily starting the second day after surgery for 7 days.

Post-operative evaluation The examiners performing clinical and radiographic assessments will be blinded to the group assignments. Follow-up appointments will be scheduled throughout the first week, as well as at 3 months and 6 months postoperatively. During each visit, the following parameters will be evaluated:

1. Clinical Assessments:

   Probing depth and bleeding index measurements will be recorded at baseline and 6 months to assess peri-implant soft tissue healing. Pain levels will be assessed using a Visual Analog Scale (VAS) on the 1st, 3rd and 7th days postoperatively.
2. Radiographic Assessment:

Cone beam computed tomography (CBCT) will be taken at (baseline) before immediate implant placement (IIP) to assess the thickness of the labial plate of bone and the patients will be exposed to another CBCT after 6 months after implant placement for evaluation of the changes in the thickness of the labial plate of bone. Readings of bone thickness will measured at three different levels: implant platform(T0), 2mm (T1) and (T2) 4mm And crestal bone loss or marginal bone loss. Statistical analysis The data will be analyzed and visualized using SAS JMP statistical software version 17.2. Descriptive statistics will be presented as mean ± standard deviation. To compare outcomes between the control and study groups at each individual time point, independent Student's T-tests will be performed. Each time point will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 1- Patients ages more than 18 years old, Participants were chosen according to specific eligibility criteria, requiring them to be healthy individuals classified as ASA I by the American Society of Anesthesiologists.

  2- Patients requiring extraction of posterior teeth with consequent immediate implant placement.

  3- Indications for extraction included: non restorable teeth (posterior teeth), untreatable caries, endodontic failures, remaining roots, vertical fracture of the roots.

  4- Natural teeth adjacent to the tooth to be extracted will required to have complete occlusal surfaces and be free from infections..

  5. Patients will selected with a thick soft tissue phenotype and a minimum keratinized tissue width (KTW) of 2 mm.

Exclusion Criteria:

* Pathologies or drugs that alter tissue integration with dental implants. 2- Head and neck radiation therapy. 3- Renal disease, bleeding disorders and anticoagulant therapy. 4- Pregnant females. 5- Patients with severe para-functional habits and unfavorable occlusion 6- Smokers. 7- Malaligned teeth and teeth with acute periapical pathosis.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
primary stability | 0, 3 months
  Evaluate the primary stability by osstell pre- and post-3-month during abutment placement, this meaure from 1-99 ISQ

SECONDARY OUTCOMES:
secondary outcomes | baseline, 3 months, and 6 months
  evaluate amount of bone gain around implant measured by CBCT this measured by mm on CBCT
secondary outcome | 3 months and 6 months
  clinical periodontal parameters (CAL, PD, and BOP), which were measured using periodontal probe by mm

CONTACTS AND LOCATIONS:
Overall Officials: aya kamal, Principal Investigator — lecturer of periodontology Minia University

IPD SHARING:
Plan to Share IPD: Undecided